CLINICAL TRIAL: NCT01085305
Title: The Effectiveness of Parent-Child Interaction Therapy (PCIT) in Treating Behavior Problems in Young Children
Brief Title: The Effectiveness of Parent-Child Interaction Therapy (PCIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2006.789
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Behavior Problems; Oppositional Defiant Disorder; Conduct Disorder
Keywords: Behavior problems; Parent-Child Interaction; Locus of control; Psychiatric symptoms; Depressive symptoms; Attachment
MeSH Terms: conditions — Mental Disorders; Oppositional Defiant Disorder; Conduct Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCIT (Experimental): Provision of Parent-Child Interaction Therapy
  Interventions: Behavioral: Parent-Child Interaction Therapy
- TAU (Active Comparator): Treatment as usual from other therapists in the same clinics
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy — Parents will be trained in interaction with their children in ways which foster non-hostility and cooperation in their children. By means of an ear-plug they will receive instruction on how to play and set limits for their child from their therapist who watches the interaction through a one-way mirror. Treatment is given until the parent masters these skill, which commonly takes 15-20 session of 1 hour.
  Arms: PCIT
Behavioral: TAU — Usual treatment for behavioral disorders
  Arms: TAU

SUMMARY:
The purpose of this study was to investigate whether a type of parent-based intervention, Parent-Child Interaction Therapy will lower symptoms of behavior problems in young children more than treatment as usual.

DETAILED DESCRIPTION:
Behaviour problems, i.e. symptoms of oppositional defiant disorder (ODD) and conduct disorder (CD) are among the prevalent psychiatric disorders in children and one of the leading causes of help-seeking for mental health problems in children. There are several efficacious treatments for such problems in young children. However, most of these require that parents meet in groups. This is not always feasible. It is therefore a need to develop treatments that can deal with parents and families individually. Parent-Child Interaction Therapy (PCIT) is such an individually based treatment. Efficacy studies indicate symptom reduction greater that in treatment as usual (TAU). However, there is a need to study its effectiveness in ordinary clinical practise. This trial will study its effect in ordinary psychiatric clinics in the middle of Norway and compare it to the regular treatment (TAU) provided to young children with behavior problems in these clinics.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Child mental health specialty clinic for behavioral or attentional/hyperactive problems
* ECBI score of > 120
* 2 to 7 years of age
* Parental consent to the study

Exclusion Criteria:

* Psychosis or serious drug abuse in parents
* Lack of sufficient proficiency in Norwegian to fill in the questionnaires
* Mental retardation or pervasive developmental disorder in the child
* Suspicion of parental neglect or abuse of the child warranting a report to the child protection services

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2006-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | Pre intervention, 6 months, 18 months
  ECBI is taken at study entry, after 6 months and after 18 months

SECONDARY OUTCOMES:
Dyadic Parent-Child Interaction Coding System (DPICS) | Pre intervention, 6 months, 18 months
  Parent-child interaction coded from standardized situations
Parenting Stress Index | Pre intervention, 6 months, 18 months
  Number and degree of perceived stresses by parents
Working Model of the Child Interview (WMCI) | Pre intervention, 6 months, 18 months
  Parents' attachment to the child
Child Behavior Check List (CBCL)/Teacher Report Form (TRF) | Pre intervention, 6 months, 18 months
  Psychiatric symptoms as rated by parents and teachers, respectively
Beck Depression Inventory (BDI) | Pre intervention, 6 months, 18 months
  Depressive symptoms in parents
Parental Locus of Control - Short Form (PLOC-SF) | Pre intervention, 6 months, 18 months
  Parents' perceptions of internal versus external locus of control

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wichstrøm, prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - barne- og ungdomspsykiatrisk klinikk, Helse Midt-Norge, Trondheim, Sør-trøndelag
  - Barne- og ungdomspsykiatrisk klinikk, Sør-Trøndelag, Trondheim, Trondheim

REFERENCES:
- [Result] Bjorseth A, Wichstrom L. Effectiveness of Parent-Child Interaction Therapy (PCIT) in the Treatment of Young Children's Behavior Problems. A Randomized Controlled Study. PLoS One. 2016 Sep 13;11(9):e0159845. doi: 10.1371/journal.pone.0159845. eCollection 2016. PMID 27622458